CLINICAL TRIAL: NCT02798055
Title: A National, Observational, Multi-center Registry to Examine the Characteristics of Patients With Systematic Sclerosis Digital Ulcers and Assess Bosentan Treatment.
Brief Title: Bosentan Treatment of Digital Ulcers Related to Systemic Sclerosis
Acronym: GRegistry SCDU
Status: Completed | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2016-BSN-EL-64
Record Dates: First submitted 2016-06-03; First posted 2016-06-14 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2018-12

CONDITIONS: Systematic Sclerosis; Digital Ulcer; Scleroderma
MeSH Terms: conditions — digital ulcers; Scleroderma, Diffuse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Bosentan group

SUMMARY:
GRegistry is a significant collection of data and information on the clinical practice of systemic scleroderma finger ulcers.

The GRegistry study is a nationwide (Greece) prospective study recording, which includes consecutive patients with SC-DU diagnosis in clinical management departments of different hospitals, selected in such a way as to reflect a representation of the country.

The use of Bosentan in the treatment of patients suffering from systemic sclerosis with digital ulcer disease is supported by data from large, placebo-controlled, randomized studies. The beneficial effect of Bosentan in digital ulcers, a vascular event of systemic sclerosis consistent with its beneficial effect on pulmonary arterial hypertension associated with connective tissue disease and its beneficial effect on vascular remodeling.

DETAILED DESCRIPTION:
The existence and use of Patient Registries, represents one of the foundations of the progressing medical science, both for studying the natural history of diseases as well as to critically evaluate the therapeutic methods, the collection and analysis of the data from a large number of hospital units, is essential. Furthermore, the assessment of the effectiveness and adequacy of health services should be based on long-term monitoring of large groups of patients, and the assessment of the efficient functioning of the individual units, is only possible only with the availability of information for the patients of these units.

Moreover, the record of health services distribution data is a prerequisite for the design of their future development. The above led to growth of many national and international patient logs, diseases and specific treatments, the operation of which has contributed to the advancement of medical science.

Scleroderma or Systemic Sclerosis (SC) is a chronic autoimmune disease of the connective tissue with an incidence of 1: 10000- 1: 30000. In Greece it is estimated that there are approximately 2,500 patients. The disease usually affects women aged 40-60 years, and the incidence is four women to one man. The pathogenesis of the disease is unknown, while the main causes are considered genetic and environmental factors.

Two of the most critical complications of the disease, are the Pulmonary Arterial Hypertension, which occurs in patients with SC approximately 8-12% of patients, being the main cause of death, and digital ulcers that occur in 30-60 % of patients and are painful sores on the fingers. Digital ulcers, i.e. painful sores on the fingers, as a consequence of the limited blood supply of vessels are seen in approximately 30-60 % of patients with scleroderma. The digital ulcers adversely affect the quality of life of patients, even the simple daily activities and can lead to serious complications, such as amputation. The symptoms of scleroderma can vary between patients and may not be typical of this disease, at least in the early stages, making it difficult to diagnose. Two of the early symptoms are disturbance of blood supply to the extremities by a color change of the skin of the fingers, alternately pallor-cyanation-redness (Raynaud phenomenon) and rigid edematous fingers.

ELIGIBILITY:
Inclusion Criteria:

* Both genders >18 and < 80 years
* ACR 2013 criteria >9 & =9
* At least one Digital Ulcer
* Raynaud Severity Scale (0-10)

Exclusion Criteria:

* < 18 years
* ACR 2013 criteria <9

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Digital Ulcers caused by Systematic Scleroderma according to ACR 2013 criteria
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Reynaud Severity Scale | 4 months
Number of Ulcers | 4 months
Modified Rodnan Skin Score - MRSS | 4 months
Complications of systems | 4 months
  Number of organic systems which are affected by Systematic Scleroderma within last 4 months

SECONDARY OUTCOMES:
Adverse Events | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic, Laiko Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided